CLINICAL TRIAL: NCT04560205
Title: Tocilizumab: A Therapeutic Cache Against the Treatment of Severe Cases of COVID-19
Brief Title: Tocilizumab in COVID-19 Lahore General Hospital
Acronym: TC19LGH
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lahore General Hospital (Other Government)
Responsible Party: Principal Investigator, Dr. M.Irfan Malik, Associate Professor of Pulmonology / Focal Person COVID-19, Lahore General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LGH001
Record Dates: First submitted 2020-07-11; First posted 2020-09-23 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: SARS-CoV Infection
Keywords: COVID-19; IL-6 Inhibitor
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19 | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: quasi-experimental
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group intervene with Tocilizumab (Experimental): Review effect of Tocilizumab as clinical trial among hospitalized patients with COVID-19 infection.
  Participants with severe disease will receive an intravenous (IV) injection of 8 mg/kg (not to exceed 800 mg) tocilizumab. Specifically, we will test whether tocilizumab is associated with a reduction in multi-organ dysfunction among hospitalized COVID-19 adult patients with elevated inflammatory biomarkers.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — 4-8mg/kg with 400mg maximum dose of Tocilizumab will be given in 60 minutes I/V infusion, and dose will be repeated after 12-24 hours according to clinical as well as laboratory parameters.
  Customized decision for Tocilizumab usage will be made by attending infectious diseases physician, comfort with Tocilizumab usage, bacterial co-infection and duration of Ventilation.
  Other Names: ACTEMRA®

SUMMARY:
The most accepted description of severe COVID-19 disease is development and over production of pro-inflammatory cytokines. Autopsy studies have been done on COVID-19 patients proved that severe disease is resulted due to deviant host-immune response and cytokine storm. Elevated inflammatory biomarkers like C-Reactive protein (CRP) and pro-inflammatory cytokines shown to be higher in severe disease of COVID-19. Several studies on severe COVID-19 have revealed raised levels of plasma cytokines like IL-6, IL-2, IL-10, Gamma interferon (INF), Tumor necrosis factor Alpha TNF. The Cytokines release syndrome (CRS) is a hyperinflammatory deadly syndrome characterized by release of uncontrolled immune system activation which is responsible for multi-organ failure. It has the main role in ARDS due to SARS-CoV-2 virus which binds to alveolar epithelium and resulting in IL-6 release that is responsible for increase alveolar-epithelium permeability. In many studies it has been observed that IL-6 have played a main role in CRS induction. Previous experiences from hyperinflammatory and cytokine storm syndromes recommends that early involvement of inhibiting CRS is essential to prevent lethal tissue damage and poor clinical outcome. In this scenario the judgement of clinical specialist who are suggesting that evidence of CRS can be cured with glucocorticoids, I/V immunoglobulin and anti-cytokine therapy cannot be ignored.

DETAILED DESCRIPTION:
This is intervention single-center study, that will be done at Lahore General Hospital in which 95 beds are allocated for COVID-19 patients including ICUs and HDUs. Ethical approval will be obtained from research ethical committee of Lahore General hospital, Lahore. Informed consent will be obtained from all patients who will agree to publish their data in this research. Patient's privacy and obey will be protected with the Helsinki Declaration.

ELIGIBILITY:
Inclusion Criteria:

* All patients of all ages, males and non-pregnant females who will be diagnosed COVID-19 positive by RT-PCR.
* Patients having classical radiological lesions of COVID-19 on X-ray chest or HRCT chest.
* Patient >55 years of age Or Age <55 with comorbid condition who will be unable to maintain O2 sat > 93% with 5-7 liter of oxygen.
* Or Patient < 55 with no comorbid conditions, who will be unable to maintain O2 sat > 93% with 7-10 liter of oxygen.
* Respiratory rate > 30-35/ min and >50% of radiological involvement of lung with typical lesions.
* Along with > 50% deranged ≥ 2 biochemical markers CRP > 50 mg/l, LDH > 1000U/L, D.Dimer > 1mg/l or 1000 ng/ml, Serum Ferritin > 1000 ng/ml or mcg/l will be included in clinical trial.

Exclusion Criteria:

* Patient who will not require supplemental oxygen during hospital stay.
* Patients on Invasive mechanical ventilation (IMV).
* Patients with respiratory rate < 30/mins and whose laboratory findings will not be deranged > 50%.
* Patients with improving radiological findings will be excluded.
* Patients suffering from Active TB
* Herpes zoster
* Multiple sclerosis,
* Allergic to tocilizumab
* Presences of chronic renal failure > 4 stage, GFR < 30ml/min/1.73m2.
* ALT/AST > 5 times than normal values.
* Presences of neutropenia < 500/mm3.
* Platelets count less than 50 ×103 /µl.
* Complicated diverticulitis/ intestinal perforation.
* Immune-suppressive anti- rejection therapy.
* Pregnant women.
* Previous MI/ IHD, IV heart failure.
* Psychiatric patients.

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical response after administration | 10 days
  Clinical improvement of COVID-19 patients by Tocillzumab The number of intubated patients. The number of patients with death.

SECONDARY OUTCOMES:
Clinical response to treatment | 15 days
  Overall survival of COVID-19 patients after drug administration.
Duration of hospitalization | 15 days
  Number of days of hospital admission either in ICU or HDUs till date of discharge
Clinical outcome of the treatment | 15 days
  Mortality rate
Supplemental Oxygen Requirement from Baseline | 15 days
  Duration of increased supplemental oxygen requirement from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Sardar Al-Fareed Zafar, Study Director — Post-Graduate Medical Institute, Lahore General Hospital, Lahore Pakistan
Locations (1):
- Lahore General Hospital, Lahore, Punjab Province, Pakistan

REFERENCES:
- [Background] Wichmann D, Sperhake JP, Lutgehetmann M, Steurer S, Edler C, Heinemann A, Heinrich F, Mushumba H, Kniep I, Schroder AS, Burdelski C, de Heer G, Nierhaus A, Frings D, Pfefferle S, Becker H, Bredereke-Wiedling H, de Weerth A, Paschen HR, Sheikhzadeh-Eggers S, Stang A, Schmiedel S, Bokemeyer C, Addo MM, Aepfelbacher M, Puschel K, Kluge S. Autopsy Findings and Venous Thromboembolism in Patients With COVID-19: A Prospective Cohort Study. Ann Intern Med. 2020 Aug 18;173(4):268-277. doi: 10.7326/M20-2003. Epub 2020 May 6. PMID 32374815
- [Background] Ramos-Casals M, Brito-Zeron P, Lopez-Guillermo A, Khamashta MA, Bosch X. Adult haemophagocytic syndrome. Lancet. 2014 Apr 26;383(9927):1503-1516. doi: 10.1016/S0140-6736(13)61048-X. Epub 2013 Nov 27. PMID 24290661
- [Background] Radbel J, Narayanan N, Bhatt PJ. Use of Tocilizumab for COVID-19-Induced Cytokine Release Syndrome: A Cautionary Case Report. Chest. 2020 Jul;158(1):e15-e19. doi: 10.1016/j.chest.2020.04.024. Epub 2020 Apr 25. PMID 32343968
- [Background] Liu B, Li M, Zhou Z, Guan X, Xiang Y. Can we use interleukin-6 (IL-6) blockade for coronavirus disease 2019 (COVID-19)-induced cytokine release syndrome (CRS)? J Autoimmun. 2020 Jul;111:102452. doi: 10.1016/j.jaut.2020.102452. Epub 2020 Apr 10. PMID 32291137
- [Background] Henderson LA, Canna SW, Schulert GS, Volpi S, Lee PY, Kernan KF, Caricchio R, Mahmud S, Hazen MM, Halyabar O, Hoyt KJ, Han J, Grom AA, Gattorno M, Ravelli A, De Benedetti F, Behrens EM, Cron RQ, Nigrovic PA. On the Alert for Cytokine Storm: Immunopathology in COVID-19. Arthritis Rheumatol. 2020 Jul;72(7):1059-1063. doi: 10.1002/art.41285. Epub 2020 May 10. PMID 32293098